CLINICAL TRIAL: NCT06422286
Title: Efficacy of Low-level Laser Acupuncture and Microcurrent Electrical Stimulation on Gag Reflex on Children During Taking Dental Impression
Brief Title: Efficacy of Low-level Laser Acupuncture and Microcurrent Electrical Stimulation on Gag Reflex on Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Baraka, Lecturer, Pediatric dentistry department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0800_11/2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Gagging
Keywords: gag reflex; dental anxiety; low-level laser
MeSH Terms: conditions — Gagging | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- children allocated to low-level laser (Experimental): The laser device with wavelength 940 nm, energy 4J, and 3-4 mm away from the tissue is applied on PC6 acupoint without causing pain to the patient for 1 minute.
  Immediately after the laser acupuncture, an alginate impression is going to be taken.
  Interventions: Device: low-level laser
- children allocated to microcurrent electrical stimulation (Experimental): A meridian acupuncture pen with AA battery will be applied on PC6 for one minute.
  Immediately after using the meridian pen, an alginate impression is going to be taken.
  Interventions: Biological: microcurrent stimulation
- placebo control group (Placebo Comparator): A meridian acupuncture pen will be deactivated by the operator. Then an alginate impression is going to be taken.
  Interventions: Device: placebo

INTERVENTIONS:
Device: low-level laser — children will be allocated to the device then the gag reflex will be re-evaluated
  Arms: children allocated to low-level laser
Biological: microcurrent stimulation — children will be allocated to the device then the gag reflex will be re-evaluated
  Other Names: meridian pen
  Arms: children allocated to microcurrent electrical stimulation
Device: placebo — children will be allocated to a deactivated meridian pen
  Arms: placebo control group

SUMMARY:
the aim of the current study is to evaluate the effectiveness of the laser acupuncture in comparison to the electroacupuncure for controlling gag reflex in children

DETAILED DESCRIPTION:
the study will select children who are suffering from gag reflex that can affect their dental appointments negatively. they will be diagnosed then randomly distributed to one of the 3 groups of the study gag reflex and anxiety will be measured before and after the intervention then the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* children free of any systemic disease or special health care needs
* children with score 2 or 3 according to the frankle behavioral rating scale
* a full arch maxillary alginate impression is needed
* moderate to severe gagging according to the gagging severity index
* written informed consent of the legal guardian

Exclusion Criteria:

* children taking anti-emetic drugs
* children sensitive to alginate

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-08-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
gagging prevetive index | immediately after the intervention
  the difference in gagging preventive index before and after the intervention

SECONDARY OUTCOMES:
anxiety | immediately after the intervention
  dental anxiety will be measured before and after the intervention using pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: sawsan hafez, PHD, Study Chair — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Baraka M, Zeitoun SI, Salah S, Hafez S. Comparative efficacy of laser and electroacupuncture on anxiety management and salivary alpha-amylase levels in pediatric dental patients with excessive gag reflexes: a randomized clinical trial. BMC Oral Health. 2025 Jul 26;25(1):1254. doi: 10.1186/s12903-025-06630-x. PMID 40713587
- [Derived] Salah S, Hafez S, Baraka M. Effect of Low-Level Laser Acupuncture and Microcurrent Electrical Stimulation on Gag Reflex in Children During Dental Impression: A Randomized Controlled Clinical Trial. Int J Paediatr Dent. 2025 Jul;35(4):848-856. doi: 10.1111/ipd.13296. Epub 2025 Jan 23. PMID 39846139